CLINICAL TRIAL: NCT02977260
Title: The Lunch Study: the Combined Effects of Food Texture and Energy Density on Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Keri McCrickerd, Dr Keri McCrickerd, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015/00867 Part 1
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Satiation
Keywords: Meal size

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Test Meal 1 (Experimental): Thin/Low Energy
  Interventions: Other: Thin/Low Energy
- Test Meal 2 (Experimental): Thin/High Energy
  Interventions: Other: Thin/High Energy
- Test Meal 3 (Experimental): Thick/Low Energy
  Interventions: Other: Thick/Low Energy
- Test Meal 4 (Experimental): Thick/High Energy
  Interventions: Other: Thick/High Energy

INTERVENTIONS:
Other: Thin/Low Energy — Thin textured rice meal (ground rice grains) with lower energy density (0.57 kcal/g)
  Arms: Test Meal 1
Other: Thin/High Energy — Thin textured rice meal (ground rice grains) with higher energy density (1.01 kcal/g)
  Arms: Test Meal 2
Other: Thick/Low Energy — Thicker textured rice meal (whole rice grains) with lower energy density (0.57 kcal/g)
  Arms: Test Meal 3
Other: Thick/High Energy — Thicker textured rice meal (whole rice grains) and high energy density (1.01 kcal/g)
  Arms: Test Meal 4

SUMMARY:
Meal size is strongly influenced by a number of external features of the food environment which can promote over-consumption, such as the availability of palatable energy dense foods. The current research aimed to investigate whether natural food-based differences in texture could be used to slow down eating rate and reduce intake from large portions and higher energy dense foods.

A four-session randomised crossover study assessed the effect of faster vs. slower eating rate, achieved through manipulating food texture, on ad-libitum consumption (weight and calories) at a meal, alone and in combination with variations in meal energy-density (higher vs. lower)

DETAILED DESCRIPTION:
The current obesogenic environment is characterized by the abundance of palatable and high energy dense foods. High dietary energy density can promote sustained overcompensation at meal times. On the other hand, eating at a slower rate has been shown to reduce meal size, and food-based texture differences can slow eating rate. It is possible that texture-based differences in eating rate could be used to reduce energy intake in of foods that are higher in energy density.

This study was conducted to quantify the effect of eating rate (fast vs. slow) on ad-libitum consumption of a meal, alone and in combination with variations in meal energy-density (0.57 kcal/g vs 1.01 kcal/g). The meal combinations were as follows:

Meal 1: thin/0.57 kcal; Meal 2: thin/1.01 kcal/g; Meal 3: thick/ 0.57 kcal/g; Meal 4: thick /1.01 kcal/g

Participants consumed the four test meals over four non-consecutive test sessions at the Clinical Nutrition Research Centre, with at least three days washout between each session. Each part followed a completely randomised full crossover design.

The primary objective was to assess ad libitum intake (both kcal and g) of the test meals, depending on the combination of food texture and energy density.

The secondary objectives were to assess the eating rate, oral processing characteristics, changes in rated appetite up to 90 minutes post-consumption and energy intake (kcal) for the rest of the test day (food diary), as a function of the test meal texture and energy density

ELIGIBILITY:
Inclusion criteria:

* Aged between 21 and 50 years
* BMI < 30 kg/m2

Exclusion criteria:

* Individuals whose body weight has changed more than 5 kilograms in the last 12 months
* People who are taking insulin or medications known to affect glucose metabolism, appetite or energy metabolism
* Individuals who are currently dieting
* People with intolerances or allergies to study foods or test products, e.g. soya, wheat, gluten, cereal, fruits, biscuits, dairy products, rice, vegetable, meat, seafood, sugar and sweetener, gelatin, natural food colourings or flavourings, etc
* Pregnant women

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Ad libitum intake of the test meals - weight (g) | Measured once for up to 20 minutes
  The weight of the test meal consumed during the test session was measured.
  There are four test sessions and participants eat one of the four test meals each session. The amount consumed was measured each time.
Ad libitum intake of the test meals - calories (kcal) | Measured once for up to 20 minutes
  The weight of the meal consumed was measured and convert to calories using the meal energy density (which is known).
  There are four test sessions and participants eat one of the four test meals each session. The amount consumed was measured each time.

SECONDARY OUTCOMES:
Eating rate of the test meals | Measured once for up to 20 minutes
  Video recordings of the participants eating are coded and from this eating rate was calculated as grams consumed per minute (g/min).
Changes in rated appetite pre- to post meal consumption and up to 90 minutes post-consumption | pre-meal, immediately post-meal, +15 minutes, +30 minutes, +45 minutes, +60 minutes, +75 minutes, + 90 minutes
  100-point Visual Analogue Scale (VAS) ratings of hunger, fullness, desire to eat, prospective consumption and thirst
Energy intake (kcal) for the rest of the test day recorded in a Food diary | Up to 24 hours
  Food intake recorded in a food diary

CONTACTS AND LOCATIONS:
Overall Officials: Keri McCrickerd, PhD, Principal Investigator — Clinical Nutrition Research Centre
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No